CLINICAL TRIAL: NCT06226519
Title: Integrated PET/MRI and Germline Variants to Differentiate Brain Tumopr Recurrence From Iatrogenicchanges in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: PET/RMN
Record Dates: First submitted 2024-01-04; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Pediatric Brain Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 11C-MET-PET/RMN — 60 children and/or adolescents (≤18 years) with a diagnosis of brain tumor (medulloblastoma, other embryonal tumors or high-grade gliomas), who have followed the contemporary adjuvant therapy protocol of post-surgical chemo and radiotherapy and completed radiotherapy for at least 6 months will undergo a brain MET-PET/MRI.

SUMMARY:
Nuclear magnetic resonance imaging (NMR) is used in pediatric brain tumors for purposes of diagnosis, evaluation of response to treatments, and monitoring of patients in follow-up. Through conventional imaging techniques it remains difficult to differentiate tumor recurrence from pseudo-progression or other iatrogenic changes after radiotherapy or chemotherapy, but it remains a relevant and essential clinical need for patient management.

ELIGIBILITY:
Inclusion Criteria:

* children and/or adolescents (≤18 years) diagnosed with brain tumor.
* children who underwent the contemporary adjuvant therapy protocol of post-surgical chemo and radiotherapy.

Exclusion Criteria:

* patients >18 years

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: 60 children and/or adolescents (≤18 years) with a diagnosis of brain tumor (medulloblastoma, other embryonal tumors or high-grade gliomas), who have followed the contemporary adjuvant therapy protocol of post-surgical chemo and radiotherapy and completed radiotherapy for at at least 6 months will undergo a brain MET-PET/MRI.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-05-13 (Actual); Primary Completion 2024-05-13 (Estimated); Study Completion 2024-05-13 (Estimated)

PRIMARY OUTCOMES:
MET-PET/brain MRI in children with brain tumor for diagnosis of brain tumor recurrence compared to therapy-induced changes. | 4 years
  The role of MET-PET/MRI and radiogenomics could play in the follow-up management of children and adolescents with brain tumors and in ensuring timely intervention in case of tumor recurrence/progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs San Raffaele, Milan, Italy